CLINICAL TRIAL: NCT05402384
Title: Evaluation of Efficacy and Safety of D-galactose Supplementation in SLC35A2-CDG, a Disorder of Hypogalactosylation
Brief Title: AVTX-801 D-galactose Supplementation in SLC35A2-CDG
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eva Morava-Kozicz (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Rare Diseases Clinical Research Network (Network); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor-Investigator, Eva Morava-Kozicz, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-005271; U54NS115198 (NIH)
Record Dates: First submitted 2022-05-28; First posted 2022-06-02 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: SLC35A2-CDG - Solute Carrier Family 35 Member A2 Congenital Disorder of Glycosylation
MeSH Terms: interventions — Galactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AVTX-801, then Placebo (Experimental): Each treatment period is 24 weeks, with 6-week washout period in between.
  Interventions: Drug: AVTX-801; Drug: Placebo
- Placebo, then AVTX-801 (Placebo Comparator): Each treatment period is 24 weeks, with 6-week washout period in between.
  Interventions: Drug: AVTX-801; Drug: Placebo

INTERVENTIONS:
Drug: AVTX-801 — Medical grade D-galactose
  dosage:2.0 g/kg/day
  Other Names: D-Galactose
Drug: Placebo — Matching placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, cross-over study to evaluate the efficacy and safety of AVTX-801 in subjects with SLC35A2-CDG

ELIGIBILITY:
Inclusion Criteria

* Molecular confirmation of SLC35A2 genetic variant
* Age > 1 month
* Presence of seizures, chronic vomiting, chronic constipation, or chronic diarrhea
* A parent or legal guardian must be available and willing to provide consent on behalf of minor subjects or adult subjects who are unable to give informed consent due to developmental disabilities.
* Use of contraception in females > age 8 years
* Previously performed eye exam within last year

Exclusion Criteria

* Aldolase-B deficiency
* Galactosemia
* Hemolytic uremic syndrome
* Hemoglobin < 7 mg/dL
* LFTs > 3x ULN
* Previously experienced severe AEs from oral galactose (severe diarrhea, vomiting, constipation, galactosuria, or increased liver glycogen storage)
* Other history of galactose intolerance as determined by the investigator
* Currently treated with ketogenic diet
* Current enrollment in another trial involving investigational compounds
* Ongoing dietary D-galactose supplementation
* Use of investigational compounds
* Pregnancy

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of major motor seizure frequency | 28 days
  Seizure burden assessed by change from baseline in 28-day major motor seizure frequency
Number of vomiting episodes | 28 days
  Vomiting frequency in 28-day from baseline
Bristol Stool Form Scale (BSFS) | average daily 28 days
  Constipation/diarrhea assessed by scale improvement toward normal stool forms from baseline in average daily 28-day Bristol Stool form scale. The BSFS classifies stool into 7 groups, type 1 (hardest) to type 7 (softest). Type 3 and Type 4 would be more indicative of normal stool.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Morava-Kozicz, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No